CLINICAL TRIAL: NCT02827253
Title: Cohort Study of Morphological Changes of the Brain by MRI in Chronic Kidney Disease Patients
Brief Title: Morphological Changes of the Brain by MRI in Chronic Kidney Disease
Acronym: KIDBRAIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Principal Investigator, Juan Manuel López Gómez, PhD, PhD, Hospital General Universitario Gregorio Marañon
Other Study IDs: HGUGM
Record Dates: First submitted 2016-06-29; First posted 2016-07-11 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis
Keywords: brain; haemodialysis; intradialytic hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Predialysis: Patients with CKD (4 and 5 stages by KDOQI guidelines) underwent MRI to obtain in vivo images of brain anatomy that were subsequently analyzed by the data processing package FreeSurfer (version 5.3). A MRI 6 months after starting haemodialysis will be performed to analyze changes in gray and white matter of the brain.
  Interventions: Device: MRI
- Haemodialysis: Patients with end stage of renal disease (ESRD) in haemodialysis underwent MRI to obtain in vivo images of brain anatomy that were subsequently analyzed by the data processing package FreeSurfer (version 5.3). A one year follow up MRI will be performed to analyze the changes in gray and white matter of the brain.
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — MRI will be performed during interdialysis period in the haemodialysis group. MRI will be performed at the beginning of the study in predialysis group.

SUMMARY:
The purpose of this study is to describe brain´s morphological changes induced by chronic kidney disease (CKD) in advanced stages (stages 4 and 5 defined by KDOQI guidelines) and also by haemodialysis using MRI.

Based on the hypothesis that hypotension may cause damage in some organs including brain the investigators study if intradialytic hypotension (IDH) causes any type of changes in gray and white matter of the brain.

DETAILED DESCRIPTION:
There will be two groups: one in haemodialysis treatment and the other with chronic kidney disease patients in advanced stages (stages 4 and 5 defined by KDOQI guidelines).

Both groups will be evaluated with a MRI without contrast. A second MRI to identify brain´s morphological changes will be performed in patients of the first group a year later and in patients of the second group that will have been begun haemodialysis six months after.

In a first transverse evaluation, eighteen haemodialysis sessions from the first group will be studied with a retrospective analysis. The first three sessions of each month for six months before the MRI will be considered.

In each session the investigators will collect haemodynamic variables (systolic arterial blood pressure pre and post dialysis), intradialytic hypotension based on different definitions (Nadir90, Nadir100, Fall20, Fall30) and proper haemodialysis variables (KtV, convective transport).

In the first group and patients with CKD that will start haemodialysis, the investigators analyse the variables considered in the transverse evaluation until complete one year follow up.

Statistical analysis will be done with SPSS version 20.

ELIGIBILITY:
Inclusion Criteria:

* Prevalent patients of haemodialysis (6 months minimum)
* Patients with CKD (stages 4 and 5)
* Informed consent signed

Exclusion Criteria:

* Refusion to participate in the study
* Presence of contraindications for MRI
* Presence of clinic neurologic disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Haemodialysis group: 2 dialysis units. Predialysis group: clinic of advanced chronic renal disease.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Morphological changes in gray matter of haemodialysis group | one year
  area (mm2), volume (mm3), mean cortical thick (mm) of each structure of brain
Morphological changes in white matter of haemodialysis group | one year
  Diffusion weighted imaging: fractional anisotropy, median diffusivity, radial diffusivity, volume ratio.
Morphological changes in gray matter of predialysis group that start haemodialysis | six months
  area (mm2), volume (mm3), mean cortical thick (mm) of each structure of brain
Morphological changes in white matter of predialysis group that start haemodialysis | six months
  Diffusion weighted imaging: fractional anisotropy, median diffusivity, radial diffusivity, volume ratio.

SECONDARY OUTCOMES:
Related factors that have influence in morphological changes in haemodialysis group | one year
  age (years), time in dialysis (months), time of treatment (hours), KtV, convective transport (L/session), anemia (hemoglobin, index resistance erythropoietin), inflammation (PCR), intradialytic hypotension (Nadir90, Nadir100, Fall20, Fall30).
Related factors that have influence in morphological changes in predialysis group | six months
  age, etiology of CKD, proteinuria, blood pressure, comorbidities.

CONTACTS AND LOCATIONS:
Overall Officials: Juan M. López Gómez, PhD, Study Chair — Hospital General Universitario Gregorio Marañon; Santiago Cedeño Mora, MD, Principal Investigator — Hospital General Universitario Gregorio Marañon; Manuel Desco, PhD, Principal Investigator — Hospital General Universitario Gregorio Marañon
Locations (1):
- Hospital General Universitario Gregorio Marañon, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
publication of design of the study

REFERENCES:
- [Background] Eldehni MT, Odudu A, McIntyre CW. Randomized clinical trial of dialysate cooling and effects on brain white matter. J Am Soc Nephrol. 2015 Apr;26(4):957-65. doi: 10.1681/ASN.2013101086. Epub 2014 Sep 18. PMID 25234925
- [Background] McIntyre CW, Goldsmith DJ. Ischemic brain injury in hemodialysis patients: which is more dangerous, hypertension or intradialytic hypotension? Kidney Int. 2015 Jun;87(6):1109-15. doi: 10.1038/ki.2015.62. Epub 2015 Apr 8. PMID 25853331